CLINICAL TRIAL: NCT02627495
Title: Predicting Pain Response to Transcranial Direct Current Stimulation for Phantom Limb Pain in Limb Amputees
Status: Completed | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, MD, PhD, MPH, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P002525
Record Dates: First submitted 2015-11-16; First posted 2015-12-11 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Phantom Limb Pain
Keywords: maladaptive plasticity; Limb amputation; phantom limb pain; tDCS; non-invasive brain stimulation
MeSH Terms: conditions — Phantom Limb | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- tDCS intervention (open label) (Experimental): Subjects will undergo tDCS stimulation
  Interventions: Device: transcranial Direct Current Stimulation (tDCS): (Soterix ©)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS): (Soterix ©) — Subjects will undergo tDCS stimulation. We will use electrodes of 35cm^2, at an intensity of 2mA on the primary motor cortex contralateral to the amputated limb (or for bilateral amputees contralateral to the most painful side). The subject will undergo stimulation for 20 minutes. The subject will have 5 sessions of stimulation during a 1 week time period.

SUMMARY:
This study explores the effects transcranial Direct Current Stimulation (tDCS, Soterix ©) on Phantom Limb Pain for patients experiencing chronic phantom limb pain in open-label study design.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent to participate in the study.
2. Subject is older than 18 years.
3. 3 months of phantom limb pain (experienced regularly for at least once a week) after the amputated limb has completely healed.
4. Average pain of at least 4 on a numeric rating scale in the previous week (NRS; ranging from 0 to 10).
5. If the subject is taking any medications, dosages must be stable for at least 2 weeks prior to the enrollment of the study.

Exclusion Criteria:

1. Pregnancy or trying to become pregnant in the next 2 months.
2. History of alcohol or drug abuse within the past 6 months as self-reported.
3. Presence of the following contraindication to transcranial direct current stimulation Ferromagnetic metal in the head (e.g., plates or pins, bullets, shrapnel) Implanted head electronic medical devices (e.g., cochlear implants)
4. Head injury resulting in loss of consciousness for at least 30 min or pos-traumatic amnesia for greater than 24 hours, as self-reported
5. Unstable medical conditions (e.g. uncontrolled diabetes, uncompensated cardiac issues, heart failure or chronic obstructive pulmonary disease).
6. Uncontrolled Epilepsy
7. Suffering from severe depression (as defined by a score of >30 in the Beck Depression Inventory).*
8. History of unexplained fainting spells or loss of consciousness as self-reported during the last 2 years.
9. History of neurosurgery, as self-reported.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2021-03-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | tDCS Intervention (Open Label)
Started | 9
Completed | 5
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | tDCS Intervention (Open Label)
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (16.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Pain as Measured by the Visual Analog Scale
Description: The VAS is a common assessment used which asks subjects to self-reportedly measure their pain on a visual scale (i.e., unbearable to none). We will use a VAS to determine subjects' pain scores. Subjects will rate their pain from 0 - indicating no pain at all, to 10 - indicating the worst pain felt. This scale is also colored, from green (at 0) to red (at 10), as a visual indicator of pain.
Time Frame: Change in outcome from baseline to 2-week follow-up (after the last day of stimulation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS Intervention (Open Label)
Number analyzed (Participants) | 9
units on a scale | -1.4 (1.14)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | tDCS Intervention (Open Label)
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT02627495/Prot_SAP_000.pdf